CLINICAL TRIAL: NCT00593775
Title: The Effect of Laser Assisted Hatching in Thawing Cycles: a Prospective Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Sophie Debrock, PhD, clinical embryologist, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ML3497; ML3497 (Registry Identifier: Ethical Committee of our University hospital)
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Placenta; Implantation
Keywords: implantation rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): control group without intervention
- AH group (Active Comparator): assisted hatching performed on the embryo
  Interventions: Procedure: assisted hatching

INTERVENTIONS:
Procedure: assisted hatching — assisted hatching with laser
  Arms: AH group

SUMMARY:
The successful hatching process is a prerequisite for implantation. Freezing/thawing cycles can impair the hatching process by introducing changes in the composition of the zona pellucida. The purpose of this study is to test the hypothesis that the implantation rate per embryo and the clinical pregnancy rate per embryo transfer is higher after embryo transfer of frozen-thawed embryos with opened or thinned ZP after assisted hatching when compared to embryo transfer of frozen-thawed embryos without assisted hatching.

All patients starting a thawing cycle (with frozen embryos on d1-d2-d3-d5) can be included in this RTC study. Assisted hatching will be performed with a non-contact 1.48 diode laser system (MTG, Germany).

DETAILED DESCRIPTION:
In view of insufficient clinical evidence demonstrating the value of AH at the start of our study and in view of the need for higher implantation and LBRs in our ART programme within a series of reimbursed cycles, a prospective randomized controlled trial was performed to evaluate the effect of AH, by modified quarter laser-assisted zona thinning (mQLAZT), in our cryopreservation program. The primary aim was to test the hypothesis that the IR per embryo transferred is higher after transfer of frozen/vitrified-thawed/warmed embryos with thinned ZP after mQLAZT when compared with the transfer of frozen/vitrified-thawed/warmed embryos without mQLAZT.

ELIGIBILITY:
Inclusion Criteria:

* All patients with frozen 2pn, embryos and blastocysts who want to start an embryo thawing cycle can be included in this study.

Exclusion Criteria:

* Patients participating in the embryo reception program are excluded.

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 647 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
clinical implantation rate per embryo transferred | at 6-8 weeks of pregnancy

SECONDARY OUTCOMES:
pregnancy rate per transfer | at 14-16 days after ovulation or 17 days after the start of progesterone supplementation in a hormone replacement freeze-thaw cycle

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M D'Hooghe, MD, Study Director — UZ Leuven
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium

REFERENCES:
- [Derived] Debrock S, Peeraer K, Spiessens C, Willemen D, De Loecker P, D'Hooghe TM. The effect of modified quarter laser-assisted zona thinning on the implantation rate per embryo in frozen/vitrified-thawed/warmed embryo transfer cycles: a prospective randomized controlled trial. Hum Reprod. 2011 Aug;26(8):1997-2007. doi: 10.1093/humrep/der161. Epub 2011 Jun 8. PMID 21659315